CLINICAL TRIAL: NCT00421590
Title: A Randomized, Partially Blind, Placebo Controlled, Crossover, Single Oral Dose Study to Assess the Effect of Concomitant Antacid (Calcium Carbonate / Magnesium Hydroxide) on the Pharmacokinetics and Pharmacodynamics of SMC021 (0.8 mg Salmon Calcitonin/200 mg 5-CNAC) in Healthy Postmenopausal Women
Brief Title: Drug Interaction of SMC021 With Concomitant Antacid (Calcium Carbonate/Magnesium Hydroxide).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CSMC021C2208
Record Dates: First submitted 2007-01-11; First posted 2007-01-12 (Estimated); Last update posted 2007-06-22 (Estimated); Status verified 2007-06

CONDITIONS: Health Postmenopausal Women
Keywords: Randomized, partially blind, placebo controlled, crossover, drug interaction with concomitant antacid, pharmacokinetics, pharmacodynamics, SMC021

INTERVENTIONS:
Drug: SMC021

SUMMARY:
This study will assess the effect of concomitant antacid on the pharmacokinetics and pharmacodynamics of SMC021

ELIGIBILITY:
Inclusion Criteria:

* Healthy postmenopausal female subjects, 40 to 70 years of age, and in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening.
* At Screening, and Baseline, vital signs (systolic and diastolic blood pressure and pulse rate) will be assessed after the subject has rested for at least three (3) minutes. All blood pressure measurements at other time-points should be assessed with the subject seated, and utilizing the same arm for each determination.
* Postmenopausal women must have no regular menstrual bleeding for at least 5 years prior to inclusion or must have been surgically sterilized at least 6 months prior to screening.
* Body mass index (BMI) must be within the range of 18 to 30. Subjects must weigh at least 50 kg to participate in this study.
* Able to communicate well with the investigator, to understand and comply with the requirements of the study. Understand and sign the written informed consent.

Exclusion Criteria:

* Smokers who report cigarette use of ≥ 5 cigarette per day. Smoking will not be allowed on the days of each dosing up to the last blood sampling or the last assessment.
* Use of any prescription drugs or over-the-counter (OTC) medication (vitamins, herbal supplements, dietary supplements) started within the last month prior to screening.
* Participation in any clinical investigation within 4 weeks prior to dosing, or less than 10 times the corresponding half life of the drug taken.
* The current or previous treatment that would affect bone metabolism/remodeling.
* Donation or loss of 400 mL or more of blood within 8 weeks prior to first dosing, or longer if required by local regulation.
* Subjects with a hemoglobin level equal to or below 7.5 mmol/L at screening.
* Significant illness within two weeks prior to dosing.
* A past medical history of clinically significant ECG abnormalities or a family history grandparents, parents and siblings) of a prolonged QT-interval syndrome.
* History of autonomic dysfunction (e.g. history of fainting, orthostatic hypotension, sinus arrhythmia).
* History of acute or chronic bronchospastic disease (including asthma and chronic obstructive pulmonary disease, treated or not treated),
* History of clinically significant drug allergy or history of atopic allergy (asthma, urticaria, eczematous dermatitis). A known hypersensitivity to the study drug or drugs similar to the study drug.
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs or which may jeopardize the subject in case of participation in the study.
* Poorly controlled diabetes
* History of malignancy of any organ system within the past 5 years
* A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result.
* HIV positive
* History of drug or alcohol abuse within the 12 months prior to dosing.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38
Dates: Start 2006-10

PRIMARY OUTCOMES:
To assess the effect of concomitant antacid (calcium carbonate / magnesium hydroxide) on the pharmacokinetics and pharmacodynamics (decrease in serum CTX-I) of SMC021 (0.8 mg salmon calcitonin/200 mg 5-CNAC)

SECONDARY OUTCOMES:
To assess the tolerability of concomitantly-administered antacid and SMC021

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigative site
Locations (1):
- Novartis Investigative site, Copenhagen, Denmark